CLINICAL TRIAL: NCT00616863
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Oxcarbazapine 600 mg Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Oxcarbazepine 600 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXCA-02
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
The objective of this study was to assess the bioequivalence of a potential generic 600 mg oxcarbazepine tablet formulation with Novartis Pharmaceutical's 600 mg oxcarbazepine tablet, Trileptal, folloiwng a single 600 mg dose administered with food.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or advers response to oxcarbazepine or any other comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, two period, 7 day washout

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morrelli, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Montreal, Quebec, Canada